CLINICAL TRIAL: NCT01660932
Title: Vascular and Metabolic Effects of Omega-3 Fatty Acids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Kon Koh, professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-201103
Record Dates: First submitted 2012-08-08; First posted 2012-08-09 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2012-08

CONDITIONS: Hypertriglyceridemia
Keywords: insulin resistance
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- omega 1 (Active Comparator): omega 1 gm
  Interventions: Drug: omega
- omega 2 (Active Comparator): omega 2 gm
  Interventions: Drug: omega
- omega 4 (Active Comparator): omega 4 gm
  Interventions: Drug: omega

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: omega
  Arms: omega 1; omega 2; omega 4

SUMMARY:
The investigators hypothesize that omega does-dependently improves vascular and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* hypertriglyceridemia

Exclusion Criteria:

* overt liver disease, chronic renal failure, hypothyroidism, myopathy, uncontrolled diabetes (HbA1c > 9%), severe hypertension, stroke, acute coronary events, coronary revascularization within the preceding 3 months, or alcohol abuse

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea